CLINICAL TRIAL: NCT00219739
Title: A Phase III Prospective Randomized Comparison of Imatinib at a Dose of 400mg in Combination With Peg-Interferon-alpha2a (Peg-IFNa2a) or Cytarabine (Ara-C)Versus Imatinib at a Dose of 600mg Versus Imatinib a Dose of 400mg for Previously Untreated Chronic Myelogenous Leukemia (CML) in Chronic Phase
Brief Title: STI571 ProspectIve RandomIzed Trial: SPIRIT
Acronym: SPIRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Novartis (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIRIT
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2016-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; Imatinib; Interferon; Cytarabine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Cytarabine

ARMS (4):
- Imatinib mesylate 400 mg (Experimental)
  Interventions: Drug: Imatinib mesylate 400 mg; Drug: Imatinib mesylate 600 mg; Drug: Imatinib 400 mg + Peg-Interferon; Drug: Imatinib mesylate 400 mg + Cytarabine
- Imatinib mesylate 600 mg (Experimental)
  Interventions: Drug: Imatinib mesylate 400 mg; Drug: Imatinib mesylate 600 mg; Drug: Imatinib 400 mg + Peg-Interferon; Drug: Imatinib mesylate 400 mg + Cytarabine
- Imatinib mesylate 400 mg +Peg interferon (Experimental)
  Interventions: Drug: Imatinib mesylate 400 mg; Drug: Imatinib mesylate 600 mg; Drug: Imatinib 400 mg + Peg-Interferon; Drug: Imatinib mesylate 400 mg + Cytarabine
- Imatinib mesylate 400 mg +Cytarabine (Experimental)
  Interventions: Drug: Imatinib mesylate 400 mg; Drug: Imatinib mesylate 600 mg; Drug: Imatinib 400 mg + Peg-Interferon; Drug: Imatinib mesylate 400 mg + Cytarabine

INTERVENTIONS:
Drug: Imatinib mesylate 400 mg
Drug: Imatinib mesylate 600 mg
Drug: Imatinib 400 mg + Peg-Interferon
Drug: Imatinib mesylate 400 mg + Cytarabine

SUMMARY:
To test whether increasing the dose of imatinib or combining it with IFNalpha or ara-C increases the rate of molecular response (as measured by the decrease in BCR-ABL transcripts after 12 months of treatment) in patients with previously untreated CML in chronic phase.

To compare overall survival in a selected arm according to molecular response at 1 year from randomization with the reference arm.

DETAILED DESCRIPTION:
Imatinib at 400 mg daily has emerged as the preferred therapy for newly diagnosed CML patients who do not undergo allogeneic stem cell transplant.

A phase III randomized study, comparing imatinib at 400 mg per day to interferon plus cytarabine in newly diagnosed chronic phase CML patients enrolled 1106 patients from June 2000 to January 2001. 553 patients were randomized to each treatment. For comparative purposes, at 6 months, 75% of patients randomized to imatinib obtained a major cytogenetic response with 51% complete responses. Despite these impressive results, only a minority of patients treated with imatinib in this study achieved a molecular remission. When analyzed by log reduction in Bcr-Abl transcript levels using quantitative RT-PCR, 39% of patients achieved a 3-log reduction in Bcr-Abl levels, but only 13% and 3% achieved a 4- and 5-log reduction, respectively.2 To improve upon these results, various groups have tried higher doses of imatinib, and combinations of imatinib with interferon alpha or cytarabine. Each of these studies has used cytogenetic responses as the major endpoint.

Each of these therapies has increased toxicity as compared to 400 mg of imatinib alone and the rates of molecular remissions have not been reported.

Thus the purpose of this study is to first determine whether higher doses of imatinib or combining Imatinib with interferon or Ara-C would result in higher rates of molecular responses and if so, in better survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with Bcr-Abl positive CML in chronic phase.
* Patients within 14 weeks of diagnosis and previously untreated for CML except for hydroxyurea and/or anagrelide.
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
* ECOG performance score of 0-2
* acceptable hepatic, renal, and cardiac function
* Informed consent signed up

Exclusion Criteria:

* Depressive syndrome not controlled
* Uncontrolled medical illnesses.
* Women with childbearing potential and male patients who are unwilling or unable to use an adequate method to avoid pregancy for the entire period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2003-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival improvement

SECONDARY OUTCOMES:
Molecular response improvement at 1 year | 1 year
Hematological, cytogenetic responses improvement | 1 year
Duration of responses improvement
Survival without progression improvement
Acceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: François GUILHOT, MD, Study Chair — Department of Oncology hematology and Cell therapy, University Hospital , 86021 Poitiers - FRANCE
Locations (1):
- University Hospital, Poitiers, France

REFERENCES:
- [Derived] Bruzzoni-Giovanelli H, Gonzalez JR, Sigaux F, Villoutreix BO, Cayuela JM, Guilhot J, Preudhomme C, Guilhot F, Poyet JL, Rousselot P. Genetic polymorphisms associated with increased risk of developing chronic myelogenous leukemia. Oncotarget. 2015 Nov 3;6(34):36269-77. doi: 10.18632/oncotarget.5915. PMID 26474455
- [Derived] Delord M, Rousselot P, Cayuela JM, Sigaux F, Guilhot J, Preudhomme C, Guilhot F, Loiseau P, Raffoux E, Geromin D, Genin E, Calvo F, Bruzzoni-Giovanelli H. High imatinib dose overcomes insufficient response associated with ABCG2 haplotype in chronic myelogenous leukemia patients. Oncotarget. 2013 Oct;4(10):1582-91. doi: 10.18632/oncotarget.1050. PMID 24123600
- [Derived] Johnson-Ansah H, Guilhot J, Rousselot P, Rea D, Legros L, Rigal-Huguet F, Nicolini FE, Mahon FX, Preudhomme C, Guilhot F. Tolerability and efficacy of pegylated interferon-alpha-2a in combination with imatinib for patients with chronic-phase chronic myeloid leukemia. Cancer. 2013 Dec 15;119(24):4284-9. doi: 10.1002/cncr.28328. Epub 2013 Sep 16. PMID 24105694
- [Derived] Preudhomme C, Guilhot J, Nicolini FE, Guerci-Bresler A, Rigal-Huguet F, Maloisel F, Coiteux V, Gardembas M, Berthou C, Vekhoff A, Rea D, Jourdan E, Allard C, Delmer A, Rousselot P, Legros L, Berger M, Corm S, Etienne G, Roche-Lestienne C, Eclache V, Mahon FX, Guilhot F; SPIRIT Investigators; France Intergroupe des Leucemies Myeloides Chroniques (Fi-LMC). Imatinib plus peginterferon alfa-2a in chronic myeloid leukemia. N Engl J Med. 2010 Dec 23;363(26):2511-21. doi: 10.1056/NEJMoa1004095. PMID 21175313